CLINICAL TRIAL: NCT07025499
Title: Piloting and Evaluation of a Group Intervention for People With Psychosis Designed to Boost Access and Usage of ICT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Jaclin Whaley, Ms. Jaclin Vozza (Whaley), McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18839
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Serious Mental Illness
Keywords: Information and Communication Technology; Recovery; social connection; community participation

STUDY DESIGN:
Intervention Model Description: Pilot evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Information and Communication Technology Group Intervention (Experimental): Participants will be given access to a tablet. With this technology, participants will be invited to set personal goals related to using this technology to foster social connection and community participation. Participants will attend a group led by two occupational therapy students and an occupational therapist focused on digital literacy and how to use technology to meet their goals. In the group, participants will learn how to use their device and how to safely access various online resources and tools to support their recovery. Participants will keep their provided devices upon conclusion of the group sessions. Participants will complete quantitative outcome measures at the start and end of the group intervention. Participants will be invited to attend a semi-structured interview one month after the completion of the group about their experiences with the program.
  Interventions: Behavioral: Group ICT Intervention

INTERVENTIONS:
Behavioral: Group ICT Intervention — Participants will be given access to a tablet. With this technology, participants will be invited to set personal goals related to using this technology to foster social connection and community participation. Participants will attend a group led by two occupational therapy students and an occupational therapist focused on digital literacy and how to use technology to meet their goals. In the group, participants will learn how to use their device and how to safely access various online resources and tools to support their recovery. Participants will keep their provided devices upon conclusion of the group sessions. Participants will complete quantitative outcome measures at the start and end of the group intervention. Participants will be invited to attend a semi-structured interview one month after the completion of the group about their experiences with the program.

SUMMARY:
Participants will be given access to a tablet. With this technology, participants will be invited to set personal goals related to using this technology to foster social connection and community participation. Participants will attend a group led by two occupational therapy students and an occupational therapist focused on digital literacy and how to use technology to meet their goals. In the group, participants will learn how to use their device and how to safely access various online resources and tools to support their recovery. Participants will keep their provided devices upon conclusion of the group sessions. Participants will complete quantitative outcome measures at the start and end of the group intervention. Participants will be invited to attend a semi-structured interview one month after the completion of the group about their experiences with the program.

ELIGIBILITY:
Inclusion Criteria:

* Specific inclusion criteria for participants in this study will include being diagnosed with a psychotic disorder, living in the Hamilton area, ability to communicate in English, and having more than one episode of psychosis. Every effort will be made to recruit participants from study with HiREB approvals #17367 and #18549, as indicated in that study's previous consent form, for those that have consented to be contacted for future research.

Exclusion Criteria:

* Exclusion criteria include currently experiencing an acute psychotic episode or medical condition that would render them incapable of meaningfully participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative interviews | From end of group intervention to 3 months
  The primary outcome is what participants will share regarding their experiences with the group intervention.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | From enrolment to end of 7-week group
  Participants will write 1-3 goals regarding their access and use of technology, and rate their importance, satisfaction, and performance with these goals.
The Media and Technology Usage and Attitudes Scale (MTUAS) | From enrolment to end of 7 week group
  Participants will rate their technology usage and attitudes towards technology

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gewurtz, PhD, MScOT, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
COPM, MTUAS, qualitative interview themes
Supporting Information: Study Protocol, SAP, ICF